CLINICAL TRIAL: NCT00090818
Title: Clinical Research Core Dental Screening Protocol
Status: Completed | Type: Observational
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040267; 04-D-0267
Record Dates: First submitted 2004-09-03; First posted 2004-09-06 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-10-28

CONDITIONS: Oral Mucosal Disease
Keywords: Dental Abnormalities; Lichen Planus; Oral Mucosal Disease; Genetic Disease; Amelogensis Imperfecta; Maxillofacial Abnormalities; Craniofacial Abnormalities; Craniofacial Genetic Abnormalities
MeSH Terms: conditions — Tooth Abnormalities; Lichen Planus; Genetic Diseases, Inborn; Maxillofacial Abnormalities; Craniofacial Abnormalities

SUMMARY:
This study will screen patients for eligibility in studies sponsored by the Craniofacial Genetics Section (HCGS), the Clinical Research Core (CRC), and other branches located within the National Institute of Dental and Craniofacial Research (NIDCR). It will also evaluate patients with diseases or abnormalities of the oral cavity or craniofacial complex, or both, for future protocol development. HCGS and CRC study the natural history of oral diseases and systemic diseases that are manifested in the maxillofacial region-the upper jaw and face. Among the diseases are lichen planus, systemic lupus erythematosus, and premalignant oral leukoplakia. Researchers also study certain acquired diseases and genetic diseases. Because many of the diseases of the maxillofacial region are poorly defined, the evaluation and characterization of patients with such diseases are goals of investigation.

Patients of any age, gender, and racial and ethnic group who have oral diseases or systemic diseases of the upper jaw and face may be eligible for the study. Women of childbearing potential, or who are pregnant or lactating, may be eligible; they would undergo procedures and tests or receive medications posing a minimal risk to the fetus or child.

Participants will undergo the following procedures:

* Complete medical history and physical examination, including a thorough examination of the head and neck; detailed examination of the teeth and gums may or may not be necessary.
* Tests of blood, urine, stool; tests for pregnancy and HIV when needed; and tests for cultures, fungi, bacteria, and parasites.
* Sampling of blood and oral tissues for diagnosis, treatment response, and disease progression.
* Electrocardiogram, x-ray, and imaging procedures, including imaging of the face.

Biopsies may be performed as needed for diagnosis and to guide therapy. The type, number, location, and frequency of biopsies depend on several factors, including the nature of the disease being evaluated. Local anesthesia is typically used unless there are contraindications. Some biopsies are done with disposable, 2 to 3 mm, round, sharp metal punches. Larger excisions with the use of an appropriate blade may be necessary for proper evaluation of a patient's condition or complete removal of something that is abnormal. The risks and discomfort associated with any of the interventions include mild pain, bleeding, and infection; there may be temporary facial paralysis, bruising, and allergic reactions.

Supportive care will be given as needed, according to the patient's diagnosis, treatment, and clinical information. Disease-related or drug-related complications, or both, will be managed through collaboration with the patient's referring physician.

DETAILED DESCRIPTION:
The purpose of this clinical research protocol is twofold: 1) to screen patients for protocol eligibility for those sponsored primarily by the Craniofacial Genetics Section, the Clinical Research Core and other Branches located within the National Institute of Dental and Craniofacial Research (NIDCR) as appropriate and 2) to evaluate patients with diseases or abnormalities of the oral cavity and/or craniofacial complex for future protocol development. Patients enrolled in this protocol will be evaluated and treated according to standard procedures and therapeutic modalities. No procedures will be done for research only. Standard or experimental biochemical, genetic and proteomic tests may be conducted on tissue or blood samples collected for diagnosis. Eligible patients will be referred to appropriate NIDCR clinical research protocols for further protocol-driven diagnostic workup and therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients of any age, gender, and racial/ethnic group with oral diseases or systemic diseases with maxillofacial manifestations that are mission relevant for the Craniofacial Genetics Section, the Clinical Research Core and other branches located within the NIDCR.

Women of childbearing potential, or who are pregnant or lactating will only undergo tests and procedures, and/or receive medications for which data exists proving minimal risk to the fetus and/or child. Only diagnosis without radiographs will be performed.

EXCLUSION CRITERIA:

Patients with significant cognitive impairment.

Pregnant patients or lactating patients, if this status precludes proposed diagnostic procedures or therapies because of known untoward effects on mother and/or child.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2004-09-01; Study Completion 2010-10-28

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States